CLINICAL TRIAL: NCT00003477
Title: Phase II Study of Antineoplastons A10 and AS2-1 Infusions in Children With Visual Pathway Glioma
Brief Title: Antineoplaston Therapy in Treating Children With Visual Pathway Glioma
Acronym: VPG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066514; BC-BT-23 (Other: Burzynski Research Institute, Inc.)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2016-12-16 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Visual Pathway Glioma
Keywords: visual pathway glioma not amenable to standard therapy; visual pathway glioma not responding to standard therapy
MeSH Terms: interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Children with a visual pathway glioma, which is not amenable to standard therapy or has not responded to standard therapy, will receive Antineoplaston therapy (Atengenal + Astugenal).
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
RATIONALE: Current therapies for children with visual pathway gliomas, which are not amenable to or have not responded to standard therapy, provide limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of children with visual pathway gliomas, which are not amenable to or have not responded to standard therapy.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on children with visual pathway gliomas, which are not amenable to or have not responded to standard therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in children with visual pathway gliomas, which are not amenable to or have not responded to standard therapy, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in children with visual pathway gliomas, which are not amenable to or have not responded to standard therapy.

OVERVIEW: This is a single arm, open-label study in which children with visual pathway gliomas, which are not amenable to or have not responded to standard therapy, receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity. After 12 months, patients with a complete or partial response or with stable disease may continue treatment.

To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

PROJECTED ACCRUAL: Approximately 20-40 patients will be accrued to this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed (unless medically contraindicated) visual pathway glioma, which is not amenable to standard therapy or did not respond to standard therapy.
* Evidence of tumor by MRI scan performed within 2 weeks prior to the study entry
* Tumor must be at least 5 mm
* No brain stem tumors

PATIENT CHARACTERISTICS:

Age:

* 6 months to 17 years

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2000/mm3
* Platelet count greater than 50,000/mm3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT/SGPT no greater than 5 times upper limit of normal
* No hepatic failure

Renal:

* Creatinine no greater than 2.5 mg/dL
* No renal insufficiency
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No severe heart disease
* No uncontrolled hypertension
* No history of congestive heart failure
* No other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No severe lung disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study
* No serious active infections or fever
* No other serious concurrent disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunomodulating agents

Chemotherapy:

* At least 4 weeks since prior chemotherapy and recovered (6 weeks for nitrosoureas)
* No concurrent antineoplastic agents

Endocrine therapy:

* Concurrent corticosteroids for cerebral edema allowed (must be on stable dose for at least 1 week prior to study)

Radiotherapy:

* At least 8 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* No prior antineoplaston therapy

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 1996-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stanislaw R. Burzynski, Tomasz J. Janicki, Gregory S. Burzynski. Antineoplastons A10 and AS2-1 in the Treatment of Children with Optic Pathway Glioma: Final Report for BT-23. Cancer and Clinical Oncology 6(1): 25-35, 2017
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve patients were recruited between June1996 and May 2004. All study subjects were seen at the Burzynski Clinic in Houston TX
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 12
Completed | 8
Not Completed | 4
Not completed — Not evalauable | 4

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: Years] | 4.5 [0.6 to 16.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks. Stable Disease (SD): <50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions and no Progressive Disease, sustained for at least four weeks. Progressive Disease (PD): >=25% increase in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 8
Participants
  Complete Response | 2
  Partial Response | 2
  Stable Disease | 3
  Progressive Disease | 1

2. Secondary Outcome: Percentage of Participants Who Survived
Description: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months overall survival
Time Frame: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
Population: All study subjects receiving any Antineoplaston therapy
Measure: Number; unit: Percentage of participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 12
Percentage of participants
  6 months overall survival | 91.7
  12 months overall survival | 83.3
  24 months overall survival | 75.0
  36 months overall survival | 58.3
  48 months overall survival | 50.0
  60 months overall survival | 50.0

ADVERSE EVENTS:
Time Frame: 8 years, 2 months
Description: Adverse event data was collected through regular patient assessment and regular laboratory testing
Groups:
- Antineoplaston Therapy: Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Antineoplaston therapy (Atengenal + Astugenal): Patients with a visual pathway glioma will receive Antineoplaston therapy (Atengenal + Astugenal)
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 9/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=12)
Seizure (Nervous system disorders) | 2 — None of the seizures were related to Antineoplaston therapy.
Somnolence/depressed level of consciousness (Nervous system disorders) | 3 — None of the somnolences/depressed levels of consciousness were related to Antineoplaston therapy.
Central venous catheter infection (Infections and infestations) | 3 — None of the central venous catheter infections were related to Antineoplaton therapy.
Fever (General disorders) | 1 — The fever was not related to Antineoplaston therapy.
Vomiting (Gastrointestinal disorders) | 1 — The vomiting was not related to Antineoplaston therapy.
Hemorrhage, CNS (Nervous system disorders) | 1 — The hemorrhage, CNS, was not related to Antineoplaston therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=12)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 4
Allergic rhinitis (including sneezing, nasal stuffiness) (Immune system disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 5
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 3
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2
Central Venous Catheter Infection (Infections and infestations) | 5
Central Venous Catheter Non-functional (General disorders) | 3
Central Venous Catheter - Other (General disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 6
Fever (General disorders) | 5
Rigors/chills (General disorders) | 3
Cushingoid appearance (Endocrine disorders) | 2
Anorexia (Gastrointestinal disorders) | 2
Auditory/Ear - Other (Ear and labyrinth disorders) | 1
Platelets (Blood and lymphatic system disorders) | 1
Central Venous Catheter Pain (General disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Hot flashes/flushes (Endocrine disorders) | 1
Dehydration (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 4
Distension/bloating, abdominal (Gastrointestinal disorders) | 1
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 3
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 8
Hemorrhage, CNS (Nervous system disorders) | 1
Hemorrhage, GU: Urinary NOS (Renal and urinary disorders) | 1
Infection (documented clinically): Abdomen NOS (Infections and infestations) | 1
Infection (documented clinically): Bladder (urinary) (Infections and infestations) | 1
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 1
Infection (documented clinically): Middle ear (otitis (Infections and infestations) | 1
Infection (documented clinically): Pharynx (Infections and infestations) | 1
Infection (documented clinically): Sinus (Infections and infestations) | 2
Infection (documented clinically): Soft tissue NOS (Infections and infestations) | 1
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 3
Infection (documented clinically): Urinary tract NOS (Infections and infestations) | 1
Opportunistic infection (Infections and infestations) | 1
Viral hepatitis (Infections and infestations) | 1
Albumin, serum-low (hypoalbuminemia) (Investigations) | 1
Alkaline phosphatase (Investigations) | 2
Bicarbonate, serum-low (Investigations) | 2
Hypercholesteremia (Investigations) | 1
Hyperglycemia (Investigations) | 2
Hypernatremia (Investigations) | 7
Hypertriglyceridemia (Investigations) | 1
Hypocalcemia (Investigations) | 3
Hypokalemia (Investigations) | 10
Hypomagnesemia (Investigations) | 3
Hypoglycemia (Investigations) | 4
Hyponatremia (Investigations) | 2
Metabolic/Laboratory - Other (Investigations) | 2
Proteinuria (Investigations) | 4
SGOT (Investigations) | 2
SGPT (Investigations) | 3
Uric acid, serum-high (hyperuricemia) (Investigations) | 2
Muscle weakness: Left-sided (Musculoskeletal and connective tissue disorders) | 1
Ataxia (incoordination) (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Mood alteration (Nervous system disorders) | 2
Neuropathy: motor (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Somnolence/depressed level of consciousness (Nervous system disorders) | 8
Tremor (Nervous system disorders) | 1
Nystagmus (Eye disorders) | 1
Ocular/Visual - Other (Eye disorders) | 2
Pain: Abdomen NOS (Gastrointestinal disorders) | 2
Pain: Back (Musculoskeletal and connective tissue disorders) | 1
Pain: Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 1
Pain: Head/headache (Nervous system disorders) | 6
Pain: Joint (Musculoskeletal and connective tissue disorders) | 1
Pain: Muscle (Musculoskeletal and connective tissue disorders) | 2
Pain: Neck (Musculoskeletal and connective tissue disorders) | 1
Pain: Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No